CLINICAL TRIAL: NCT01110967
Title: Satellite™ PEEK Nucleus Replacement Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: Satellite Retrospective
Record Dates: First submitted 2010-04-15; First posted 2010-04-27 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Degenerative Disc Disease, Lumbar; Disc Herniation, Lumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Satellite™ Retrospective Analysis is an international, retrospective, multi-center, non-interventional post-marketing study designed to document and analyze existing data with the device in a "real-world" setting.

The purpose of this study is to evaluate number of adverse device effects (ADEs), serious adverse device effects (SADEs) and serious adverse event (SAEs) and early clinical effectiveness for the Satellite™ Nucleus Replacement in a standard clinical practice. Data collection will include information on health related quality of life (QoL), physical functioning and adverse event after nucleus replacement surgery. Radiographic measures will also be assessed to evaluate changes in disc height at the operated level and changes in segmental range of motion.

All patients who were implanted with a Satellite™ Nucleus Replacement Prosthesis in the participating sites are eligible for participation in the Satellite ™ Retrospective Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have signed a Patient Data Release Form
* Age of at least 18 years and skeletally mature at the time of surgery

Exclusion Criterion:

* Patient has not reached the age of legal consent according to local laws

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were implanted with a Satellite™ Nucleus Replacement device at the participating sites are eligible for participation in the Satellite ™ Retrospective Analysis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Masaryk Hospital, Ústí nad Labem, Czechia
- ÚVN SNP, Ružomberok, Slovakia
- Instituto de Columna de Caracas, Caracas, Venezuela

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Implanted With a Satellite Device
Started | 40
Surgery | 40
1 Month Follow up | 26
3 Months Follow up | 28
6 Months Follow up | 24
12 Months Follow up | 31
Completed | 31
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Region of Enrollment [Number; unit: participants]
  Czech Republic | 2
  Slovakia | 8
  Venezuela | 30

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life Using the Visual Analogue Scale for Back Pain
Description: The Visual Analogue Scale (VAS) is a tool widely used to measure pain. It is a 10 cm scale, 0cm means 'no pain' and 10cm means 'worst possible pain'. The patients mark the location corresponding to the amount of back pain they experienced on the 10cm line.
Time Frame: Up to 12 months follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 32
units on a scale
  Back pain pre-operative (n = 32) | 5.5 (2.7)
  Back pain at 1 month Follow up (n = 25) | 2.6 (2.2)
  Back pain at 3 months Follow up (n = 25) | 2.2 (2.3)
  Back pain at 6 months Follow up (n = 18) | 1.9 (1.8)
  Back pain at 12 months Follow up (n = 26) | 1.3 (1.6)

2. Primary Outcome: Health-related Quality of Life Using the Visual Analogue Scale for Leg Pain
Description: as for outcome 1
Time Frame: Up to 12 months follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 30
units on a scale
  Leg pain pre-operative (n = 30) | 7.2 (2.0)
  Leg pain at 1 month Follow up (n = 25) | 1.8 (2.1)
  Leg pain at 3 months Follow up (n = 25) | 1.0 (1.3)
  Leg pain at 6 months Follow up (n = 18) | 0.3 (0.8)
  Leg pain at 12 months Follow up (n = 26) | 0.3 (0.8)

3. Primary Outcome: Physical Functioning Using the Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) derives from the Oswestry Low Back Pain Questionnaire, it is used to measure disability for low back pain. The index is scored from 0 to 50; 0 meaning 'no disability' and 50 meaning 'maximum disability'.
Time Frame: Up to 12 months follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 38
units on a scale
  ODI pre-operative (n = 38) | 48.2 (19.6)
  ODI at 1 month Follow up (n = 26) | 23.2 (16.0)
  ODI at 3 months Follow up (n = 30) | 18.6 (12.4)
  ODI at 6 months Follow up (n = 23) | 17.5 (13.0)
  ODI at 12 months Follow up (n = 29) | 11.4 (9.2)

4. Secondary Outcome: Range of Motion (ROM) at Implanted Level
Description: The range of motion (ROM) was calculated as the angle of the segment on the flexion radiograph minus the angle of the segment on the extension radiograph, expressed in degrees (absolute value).
Time Frame: Up to 12 months follow up visit
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 22
degrees
  ROM pre-operative (n = 22) | 10.0 (7.9)
  ROM at 3 month Follow up (n = 20) | 14.3 (5.8)
  ROM at 6 month Follow up (n = 16) | 12.1 (9.8)
  ROM at 12 month Follow up (n = 16) | 14.9 (6.1)

5. Secondary Outcome: Intervertebral Disc Space (IVD) at Implanted Level
Description: The Intervertebral Disc Space (IVD) was measured as average disc height, calculated as [(A+B)/2]/H, where A is the posterior intervertebral disc height, B is the anterior intervertebral disc height and H is the anterior height of upper vertebral body.
Time Frame: Up to 12 months follow up visit
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 35
mm
  IVD pre-operative (n = 35) | 0.30 (0.08)
  IVD post-operative (n = 29) | 0.29 (0.07)
  IVD at 3 months Follow up (n = 21) | 0.28 (0.07)
  IVD at 6 months Follow up (n = 18) | 0.26 (0.06)
  IVD at 12 months Follow up (n = 19) | 0.26 (0.06)

6. Secondary Outcome: Device Subsidence Measured as Interbody Height Ratio (IBHR)
Description: Interbody Height Ratio (IBHR) is calculated as the total vertical height of the two vertebral bodies directly superior and inferior to the implant divided by the anteroposterior diameter of the superior vertebral body.
Time Frame: Up to 12 months follow up visit
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 34
ratio
  IBHR at surgery (n = 34) | 1.9 (0.2)
  IBHR at 3 months Follow up (n = 20) | 1.9 (0.2)
  IBHR at 6 months Follow up (n = 18) | 1.7 (0.2)
  IBHR at 12 months Follow up (n = 21) | 2.0 (0.7)

7. Secondary Outcome: Changes in Device Placement
Time Frame: Up to 12 months follow up visit
Measure: Number; unit: participant
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 35
participant | 1

8. Primary Outcome: Safety by Evaluating the Number of Serious Adverse Device Effects (SADEs), Adverse Device Effects (ADEs) and Serious Adverse Events (SAEs)
Time Frame: Patients were followed up according to the local practice, up to 1 year
Measure: Number; unit: events
Arm/Group | Patients Implanted With a Satellite Device
Number analyzed (Participants) | 40
events | 7

ADVERSE EVENTS:
Time Frame: Patients were followed up according to the local practice, up to 1 year
Arm/Group | Patients Implanted With a Satellite Device
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With a Satellite Device (N=40)
Residual Radiculopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Implanted With a Satellite Device (N=40)
Residual Radiculopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain and Sciatica (Musculoskeletal and connective tissue disorders) | 3 (3)
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to the retrospective design, it was not possible to report on SF-36 results and Modic endplate changes results as limited data was available in the patient records.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential Information shall not be disclosed and shall be sole property of sponsor during the term of the agreement and for 3 years after agreement termination. Results might be published or presented, however sponsor should receive publication for review at least 7 days prior to submittal. Sponsor shall limit its review to a determination of whether Confidential Information is disclosed, to allow sponsor to protect its rights in copyrightable material, and to check for technical correctness.